CLINICAL TRIAL: NCT01921595
Title: Impact of Balanced Slat Colloid HES 130/0.42 on Coagulation Profiles in Patients Undergoing Spinal Cord Tumor Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It ended early because it would not be possible to meet the target number.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4-2013-0350
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2015-12

CONDITIONS: Coagulation
Keywords: balanced salt colloid, coagulation profiles, spinal cord tumor
MeSH Terms: conditions — Thrombosis; Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valanced salt colloid group (Experimental)
  Interventions: Other: Valanced salt colloid
- Valanced salt crystalloid group (Active Comparator)
  Interventions: Other: Valanced salt crystalloid group

INTERVENTIONS:
Other: Valanced salt colloid — Maximum dose : 30ml/kg, IV, The infusion of valanced salt colloid is started at bleeding and continued until reach at maximum dose
  Arms: Valanced salt colloid group
Other: Valanced salt crystalloid group — Maximum dose : 30ml/kg, IV, The infusion of valanced salt crystalloid is started at bleeding and continued until reach at maximum dose
  Arms: Valanced salt crystalloid group

SUMMARY:
The purpose of study is to compare the effect of coagulation profile in patients receiving intraoperative balanced salt colloid undergoing spinal cord tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult patients over the age of 20 scheduled for spinal tumor removal and fixation

Exclusion Criteria:

* 1. Renal failure 2. Preexisting congestive heart failure(NYHA III ~ IV) 3. Anemia 4. Coagulopathy 5. Abnormal liver function 6. Anti coagulation/Anti platelet ,edication 7. Foreigner, illiterate 8. Disabled person,

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Compare the effect of coagulation profile in patients receiving intraoperative balanced salt colloid undergoing spinal cord tumor surgery. | up to 24hrs after anesthesia induction
  ROTEM, CBC, PT/aPTT,ABGA, Lactic acid, electrolyte

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea